CLINICAL TRIAL: NCT05313451
Title: Evaluation of the Effect of a Soluble Fiber Consumption on the Immune Response Post-influenza Vaccination in Healthy Subjects Aged 50 to 70 Years
Brief Title: Evaluation of the Effect of a Soluble Fiber Consumption on Immunity Response
Acronym: NUTIVAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEN Biotech (Industry)
Collaborators: Roquette Freres (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1699
Record Dates: First submitted 2022-03-02; First posted 2022-04-06 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-08

CONDITIONS: Immune Response

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soluble fiber (Experimental): Participants ingest 15 g daily of the experimental product for 2 months and receive the influenza vaccine at the end of the first month.
  Interventions: Other: Soluble fiber
- Placebo (Placebo Comparator): Participants ingest 15 g daily of the placebo product for 2 months and receive the influenza vaccine at the end of the first month.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Soluble fiber — 15g/day during 2 months
  Arms: Soluble fiber
Other: Placebo — Maltodextrin 15g/day during 2 months
  Arms: Placebo

SUMMARY:
At European level, the European Food Safety Agency has recognized two claims relating to the effects of prebiotics on the gastrointestinal sphere and on the immune system. In subjects aged 45-63, it was shown that a pre- and post-vaccination inulin consumption of 8g/day significantly increased the titer of antibodies directed against the H3N2 viral strain. The increase in bifidobacteria in the faeces confirmed that this effect was related to prebiotic capacities. The effect of prebiotics and probiotics on the immune response to influenza virus vaccination has been studied in two systematic reviews and meta-analyses. The authors show that the consumption of prebiotic fibers such as FOS, GOS, inulin, was also effective on the H3N2 strain, as on the H1N1 and B strains (antibody titers of 19.5%, 20.0% and 13.6% higher, respectively, compared to placebo).

The soluble fiber under study is a resistant dextrin meeting the definition of a prebiotic fibre. The prebiotic properties have been demonstrated in humans in several studies for doses ranging from 10 to 20 g/day. Similarly, studies show that the effects on immune functions are favorably impacted by a consumption of 10 g/day for 8 weeks . These results confirm those of a preclinical study conducted in mini-pigs.

The main objective of these study is to demonstrate that these prebiotic properties could help stimulate the post-vaccination immune response, and more specifically the production of antibodies directed against seasonal influenza viruses (following vaccination), and modulate the pro- and anti-inflammatory responses.

DETAILED DESCRIPTION:
Screened participants who met the eligibility criteria are randomized either in the control or test (soluble fiber) group.

They are asked to ingest placebo or test product at 15 g/d dosing for 60 days (2 months) . At the end of the first month (30 days) they get vaccinated against influenza virus. The effect of soluble fiber on immune response is assessed by the comparison of HI titration 30 days after vaccination between groups.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject with a body mass index (BMI) of 18.0-30.0 kg/m 2
* Subject with regular upper respiratory tract infections(nasopharyngitis, flu-like illness, flu, cold...)
* Subject accepting the anti-influenza virus vaccination
* Subject agreeing to maintain lifestyle and dietary habits over the study

Main Exclusion Criteria:

* Subject having had the flu during the current season
* Subject having presented a viral or bacterial infection in the past 7 days prior to inclusion
* Subject with a known allergy to one of the compounds of products administered in the study or in accordance with indications of the vaccine
* Subject having presented manifestations of allergy during previous flu vaccinations
* Subject with ongoing gastrointestinal disease or chronic gastrointestinal disease (IBS, Crohn's disease, etc.)
* Suffering from diabetes, an autoimmune disease, a disease inflammation or a major or progressive pathology
* Pregnant women (negative urine pregnancy test for women of childbearing age), breastfeeding or planning a pregnancy in the coming months
* Subject who has already received the influenza vaccine for the current season
* Subject having received any vaccination during the last month prior to inclusion
* Subject who received antibiotic therapy within the last two month
* Taking any dietary supplements or enriched foods that are presented as having an action on immunity and/or on the intestinal sphere (prebiotics, probiotics, vitamins, plant extracts...) in the last month.
* Taking immunomodulatory or immunosuppressive drugs
* Taking any treatment that the investigator believes may interfere with investigation endpoints.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline HI titers at 2 months | at Month 1 (before influenza vaccination), at Month 2 (one month after influenza vaccination)
  hemagglutination inhibition (HI) antibody titers after vaccination

SECONDARY OUTCOMES:
Intestinal Microbiota | at month 0, At month 1, at month 2
  The microbiota is characterized using the Shotgun bacterial DNA analysis method on feces samples
Inflammatory biomarker | at month 0, at month 1, at month 2
  Interleukins
Cytokin biomarker | at month 0, at month 1, at month 2
  Tumour Necrosis Factor alpha cytokin
Incidence of Treatment on hematologic blood parameters | at month 0, at month 1, at month 2
  Complete blood count
Incidence of Treatment on biochemical blood parameters | at month 0, at month 1, at month 2
  Transaminases

CONTACTS AND LOCATIONS:
Locations (1):
- CEN Nutriment, Dijon, Bourgogne-Franche-Comté, France

IPD SHARING:
Plan to Share IPD: Undecided